CLINICAL TRIAL: NCT02474654
Title: An Analysis of the Functional Benefit, Narcotic Use and Time to Discharge Readiness Following the Implementation of a Comprehensive Pain Management Protocol for Primary Total Knee Arthroplasty
Brief Title: Implementation of a Pain Management Protocol for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Health Sciences North Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-009
Record Dates: First submitted 2015-05-06; First posted 2015-06-18 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Knee Replacement, Total
MeSH Terms: interventions — Fentanyl; Saline Solution; Epinephrine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1: PI+FNB+IO (Experimental): Bupivicaine 15mg, Fentanyl 15mcg, Epimorphine 150mcg, 0.5% Ropivicaine with 1:400,000 Epinephrine 30ml, Ropivicaine 100ml, Epinephrine 600mcg, Ketorolac 30mg
  Interventions: Drug: Bupivicaine; Drug: Fentanyl; Drug: Epimorphine; Drug: Ropivicaine; Drug: Epinephrine; Drug: Ketorolac; Drug: Ropivicaine with Epinephrine
- Arm 2:NS+FNB+IO (Experimental): Bupivicaine 15mg, Fentanyl 15mcg, Epimorphine 150mcg, 0.5% Ropivicaine with1:400,000 Epinephrine 30ml, Normal Saline 100ml
  Interventions: Drug: Bupivicaine; Drug: Fentanyl; Drug: Epimorphine; Drug: Normal Saline; Drug: Ropivicaine with Epinephrine
- Arm 3: PI+NS+IO (Experimental): Bupivicaine 15mg, Fentanyl 15mcg, Epimorphine 150mcg, Normal Saline 30ml, Ropivicaine 100ml, Epinephrine 600mcg, Ketorolac 30mg
  Interventions: Drug: Bupivicaine; Drug: Fentanyl; Drug: Epimorphine; Drug: Normal Saline; Drug: Ropivicaine; Drug: Epinephrine; Drug: Ketorolac
- Arm 4: PI+FNB+NS (Experimental): Bupivicaine 15mg, Fentanyl 15mcg, Normal Saline 0.3ml, 0.5% Ropivicaine with 1:400,000 Epinephrine 30ml, Ropivicaine 100ml, Epinephrine 600mcg, Ketorolac 30mg
  Interventions: Drug: Bupivicaine; Drug: Fentanyl; Drug: Normal Saline; Drug: Ropivicaine; Drug: Epinephrine; Drug: Ketorolac; Drug: Ropivicaine with Epinephrine
- Arm 5:NS+NS+IO (Active Comparator): Bupivicaine 15mg, Fentanyl 15mcg, Epimorphine 150mcg, Normal Saline 30ml, Normal Saline 100ml
  Interventions: Drug: Bupivicaine; Drug: Fentanyl; Drug: Epimorphine; Drug: Normal Saline

INTERVENTIONS:
Drug: Bupivicaine — 15mg
Drug: Fentanyl — 15mcg
Drug: Epimorphine — 150mcg
  Arms: Arm 1: PI+FNB+IO; Arm 2:NS+FNB+IO; Arm 3: PI+NS+IO; Arm 5:NS+NS+IO
Drug: Normal Saline — 0.3 ml
  Arms: Arm 4: PI+FNB+NS
Drug: Normal Saline — 30ml
  Arms: Arm 3: PI+NS+IO; Arm 5:NS+NS+IO
Drug: Normal Saline — 100 ml
  Arms: Arm 2:NS+FNB+IO; Arm 5:NS+NS+IO
Drug: Ropivicaine — 100 ml
  Arms: Arm 1: PI+FNB+IO; Arm 3: PI+NS+IO; Arm 4: PI+FNB+NS
Drug: Epinephrine — 600 mcg
  Arms: Arm 1: PI+FNB+IO; Arm 3: PI+NS+IO; Arm 4: PI+FNB+NS
Drug: Ketorolac — 30 mg
  Arms: Arm 1: PI+FNB+IO; Arm 3: PI+NS+IO; Arm 4: PI+FNB+NS
Drug: Ropivicaine with Epinephrine — 0.5% 1:400,000 30ml
  Arms: Arm 1: PI+FNB+IO; Arm 2:NS+FNB+IO; Arm 4: PI+FNB+NS

SUMMARY:
Study question: Is there an ideal combination of intraoperative long acting analgesics (periarticular infiltration (PI), femoral nerve block (FB) and intrathecal opioids (IO)) to optimize post-operative functional recovery, decrease overall narcotic consumption and enable faster 'readiness to discharge' for patients undergoing primary total knee replacement (TKR)?

DETAILED DESCRIPTION:
Our study design is a five-arm double blinded randomized control trial. In order to create a blinded study, each participant will have all three interventions (Femoral Nerve Block (FB), Periarticular Injection (PI) and Intrathecal Opioid (IO)) performed during their visit. Normal saline (NS) will be substituted for opioid or local anesthetic in cases where a control is required.

Specific 5 arms include:

* Using all three anesthetics:

  o PI + FB + IO (arm 1)
* Using a combination of two anesthetics + normal saline substitute for control:

  * NS + FB + IO (arm 2)
  * PI + NS + IO (arm 3)
  * PI + FB + NS (arm 4)
* Control:

  * NS + NS + IO (arm 5)

The control arm would include IO as the sole intervention as this is simply added to the spinal anesthetic used for the surgery itself. It is felt that having a study arm without any long-acting analgesic medication (opioid or local anesthetic) as the "control" arm following a spinal anesthetic would not meet current standard of care and cause harm to the participant

The investigators hypothesize that the combination of three forms of long acting analgesia (PI, FB, IO) will result in the greatest outcomes compared to a combination of any two or control. Our aim is to demonstrate that this optimal analgesic combination will have an additive pain control effect and will minimize side effects thus translating to less acute pain, improve patient mobility, and attaining "readiness to discharge" quicker.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* primary total knee replacement for osteoarthritis
* agrees to a spinal anesthetic for TKR

Exclusion Criteria:

* History of chronic pain or opioid tolerance (individuals requiring equivalent of 1 mg or more intravenous or 3 mg or more oral morphine per hour for greater than 1 month)
* general anesthetic for TKR
* major neurological deficit
* allergy to local anesthetic
* allergy to morphine or hydromorphone, anti-inflammatory, acetaminophen
* renal insufficiency
* liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-07; Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Time to Discharge | Post-op day 1 to discharge date or day 5
  Meeting discharge criteria - Participants will be followed for the duration of hospital stay, approximately 3-5 days

SECONDARY OUTCOMES:
Time up and go performance measures | Post-op day1 to discharge date or day 5
  Measured by physiotherapists - Functional Outcome - Participants will be followed for the duration of hospital stay, approximately 3-5 days
Total Opioid Consumption Measures | Post-op day 0 to discharge date or day 5
  Narcotic Use and Assessment - Participants will be followed for the duration of hospital stay, approximately 3-5 days
Complications | Post-op day 0 to discharge date or day 5
  To include nausea, vomiting, pruritis as assessed by Common Terminology Criteria for Adverse Events (CTCAE) - Participants will be followed for the duration of hospital stay, approximately 3-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wong, MD, FRCPC, BSc, PT, Principal Investigator — Health Sciences North
Locations (1):
- Health Sciences North Research Institute, Greater Sudbury, Ontario, Canada